CLINICAL TRIAL: NCT00002451
Title: A Multicenter, Open-Label, 24-Week Pilot Study to Evaluate the Safety and Activity of Indinavir Sulfate 1200 Mg q.d. and Ritonavir 200 Mg q.d. in Combination With Stavudine and Lamivudine in Treatment Naive HIV-1 Infected Patients
Brief Title: Safety and Effectiveness of Giving Indinavir, Ritonavir, Stavudine, and Lamivudine to HIV-Infected Patients Who Have Never Received Anti-HIV Drugs
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 246U; 104-00
Record Dates: First submitted 2000-01-17; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-07

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Stavudine; HIV Protease Inhibitors; CD4 Lymphocyte Count; Ritonavir; Lamivudine; Indinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Ritonavir; Lamivudine; Stavudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Ritonavir
Drug: Lamivudine
Drug: Stavudine

SUMMARY:
The purpose of this study is to see if it is safe to give indinavir (IDV) and ritonavir (RTV) in combination with stavudine (d4T) and lamivudine (3TC) to HIV-positive patients who have never received anti-HIV therapy. This study will look at the effectiveness of this drug combination and side effects.

DETAILED DESCRIPTION:
Patients entering this study initiate antiretroviral therapy. For 24 weeks patients receive daily dosages of IDV, RTV, 3TC, and d4T. Patients are seen at Day 1 and at Weeks 2, 4, 8, 12, 16, 20, and 24 for physical examinations, pregnancy testing, and blood sampling to monitor CD4 count and viral load. On Day 14, blood is drawn frequently for 24 hours for IDV and RTV pharmacokinetic sampling. The incidence of serious and drug-related adverse events and of adverse events leading to study discontinuation is tabulated.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Are at least 18 years old.
* Have a viral load of 5,000 copies/ml or greater.
* Have a CD4 count of at least 50 cells/mm3.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have taken any antiretroviral (anti-HIV) agent.
* Are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Univ of Miami School of Medicine, Miami, Florida
  - Albany Med College, Albany, New York
  - SUNY at Stony Brook / Division of Infectious Diseases, Stony Brook, New York